CLINICAL TRIAL: NCT04386421
Title: A Comparison of Three Different Modalities in Improving Oral Hygiene in Adult Orthodontic Patients - A Randomized Controlled Trial
Brief Title: A Comparison of Three Different Modalities in Improving Oral Hygiene
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr. Umair Shoukat, Co-investigator, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-1506-10214.
Record Dates: First submitted 2020-05-04; First posted 2020-05-13 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Oral Disease
Keywords: fixed orthodonitcs treatment; Adult orthodontics
MeSH Terms: conditions — Mouth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- video group (Experimental): Group A: A 3 minute video will be shown providing information regarding the care of the dentition during Fixed Appliance Treatment along with the importance of patient compliance and cooperation. The video will also be showing the consequences of poorly followed instructions such as gingivitis and white spot lesions. Participants in this group will also receive the same video graphic educational material through their Whats app once weekly for a total duration of 3 months.
  Interventions: Other: Video on oral hygeine instructions
- Plaque disclosing tablet (Experimental): Group B: Plaque-disclosing tablets will be taken by patients on chair-side showing the location of the biofilm. The patients will be given plaque disclosing tablets to be used once weekly for 3 months to evaluate their oral hygiene at home. They will be given written information in the form of leaflets on importance of cooperation and compliance. Participants in this group will receive a reminder log fill, and tablets that are not used will be asked to return to the investigator by the participants to check the compliance.
  Interventions: Drug: Plaque disclosing tablets
- Control. verbal instructions (No Intervention): Control Group C: Controls will be given only routine verbal OHI and will be briefed on the importance of cooperation and compliance at every orthodontic visit for a period of 3 months study. They will receive a reminder log that they will return at the end of the study to check compliance.

INTERVENTIONS:
Other: Video on oral hygeine instructions — A 3 minute video will be shown providing information regarding the care of the dentition during Fixed appliance treatment along with the importance of patient compliance and cooperation. The video will also be showing the consequences of poorly followed instructions such as gingivitis and white spot lesions.
  Arms: video group
Drug: Plaque disclosing tablets — Plaque disclosing tablets:
  Product: 2-Tone Disclosing Tablets Young Dental Manufacturing 13705 Shoreline Court East Earth City, MO 63045 Composition: Flavor, SD Tutti Fruiti 1 %, D and C Red 1 % and FD and C Blue 1 %
  Other Names: Plaque disclosing agent
  Arms: Plaque disclosing tablet

SUMMARY:
The objective of the study is to compare effectiveness of OHI modalities a. verbal vs videographic material, b. Verbal vs plaque disclosing tablet and c. Videographic material vs plaque disclosing tablet over 3 months in adult orthodontic patients undergoing Fixed Appliance Treatment (FAT). Secondary objective of this study is to evaluate influence of three different modalities on patient cooperation and compliance towards orthodontic treatment.

DETAILED DESCRIPTION:
It has been demonstrated that a rapid decline in oral hygiene compliance occurs after the initial bonding of fixed appliances, as orthodontic brackets favor plaque accumulation by hindering routine oral hygiene procedures such as tooth brushing and flossing. Tooth brush access to the buccal surfaces of teeth becomes problematic and predisposes plaque buildup around brackets. Inefficient removal of supra-gingival plaque leads to the development of gingival inflammation and hyperplasia.

SAMPLE SIZE:

Sample size is calculated in OpenEpi (version 3.01) sample size calculator using findings of westmead who reported mean change in verbal group for BI as 0.93 ± 0.07 (Pre-instructions = 2.31 ± 0.50 and Post-instructions = 3.24 ± 0.43) and mean change in plaque disclosing tablet group for BI as 2.9±0.21 (Pre-instruction = 4.30 ± 0.46 and Post-instruction = 1.39 ± 0.25) keeping the power of test as 90% and confidence interval of 95%, the calculated sample size came out as 1 in each group. Richter et al who reported mean compliance in low adherent group of 62.2 ± 32.3 in initial leveling and alignment of orthodontic treatment and 81.4 ± 15.5 in molar correction or space closure stage. Keeping α = 0.05 and a power of 80% sample size was calculate to be 33. Therefore we will take 33 subjects in each group.

RANDOMIZATION : Permuted block Randomization with blocks of 6 will be utilized to ensure equal representation of all 3 arms in each block. The eligible subjects in each group will be randomized to one of three groups at a 1:1:1 allocation ratio. Randomization will aid in minimizing selection bias.

ALLOCATION CONCEALMENT MECHANISM Sealed opaque envelopes containing random group information will be used in this trial, thus preventing tampering and reading of the assigned group before the subject number is given. The sealed opaque envelops will be produced by the CTU department using a system that automates the random assignment of treatment arms to subject numbers with a 1:1:1 allocation ratio within each age group. Designated CTU personnel will be responsible to the production of the randomization list and the sealed envelopes. Study staff will collect the envelopes from CTU pharmacist prior to randomization. They must be stored in a secure place and opened one by one, only after the subject has been found eligible to be randomized.

SEQUENCE GENERATION The Randomization list with treatment allocation sequence will be electronically generated using a Randomization program at CTU. CTU will maintain the randomization sequence as it is not involved in recruitment, so as to ensure allocation concealment. The envelopes will be opened sequentially following subject IDs for each consented participant after confirming the eligibility criteria BLINDING: As this is an open-label study so study subjects and investigators are not blinded.

RATIONALE:

Orthodontic patients are at an increased risk of developing gingivitis and white spot lesions due to presence of arch wire and brackets, making oral hygiene maintenance difficult. These symptoms due to poor oral hygiene will depict less interest of patients towards orthodontic treatment. Decreased and poor compliance of orthodontic patients may not only affect the health but also the overall esthetic outcome of the orthodontic treatment. So, awareness regarding oral hygiene maintenance is important. Motivations and encouragement of patients to improve oral hygiene, improve cooperation and compliance of patients towards orthodontic treatment. Various means of communication has been used by authors to evaluate the improvement in oral hygiene practices such as verbal instructions, written and educational videos. The use of plaque disclosing tablet enabled subjects to remove 19% more plaque compared to brushing alone. Presenting video graphic information regarding oral hygiene practice and sequel of plaque deposition also resulted in a significant improvement in patient knowledge thus improving oral hygiene in orthodontic patients. However, none of the aforementioned modalities have been compared with each other at a time. Therefore, the aim of this study will be to compare the overall oral hygiene improvement in fixed orthodontic patients receiving Oral Hygiene Instructions in the form of verbal briefing, demonstration via plaque disclosing tablets or video graphic information. Establishing the most efficacious modality will aid in providing Oral Hygiene Instructions that are easier to understand, retain and practice in our population undergoing Fixed Appliance Treatment.

Literature studies are evident that improvement in oral hygiene by means of various incentives improved patient cooperation and compliance. In this study the investigators will also assess whether these interventions apart from its impact on oral hygiene, has any impact on compliance and cooperation of the patient as well. A positive change with these interventions will help in better patient care and good adherence of patient with Fixed Appliance Treatment.

DATA COLLECTION:

Due to ethical considerations and patients' equal rights for oral health, all groups will receive routine Oral Hygiene Instructions. The patients will be randomly allocated into 1 of the 3 groups. Data will be collected four times during the whole study from a single participant, initial baseline measurement (T0) will be taken on the first visit after inclusion in the study however second, third and fourth measurement will be taken (T1, T2, T3) after 1, 2 and 3 months follow up visits of the participant. Data for both the baseline scores and after intervention scores will entered in the designed proforma which includes all the indices used in this study

Patient cooperation will also be determined after 3 months by Orthodontic Patient Cooperation Scale (OPCS). This questionnaire will be filled by the patients' attending orthodontist. It consists of 8 questions to assess cooperation and compliance of patient. Scale covers parameters like attitude of patient towards orthodontic treatment, attitude of patient with doctor, responsible attitude of patient, interest of patient etc. Each question contains equal scores. Maximum scores being 5 and minimum 1. Percentage of scores will be calculated. Total Scores below 34% will be considered as low cooperation, while scores ranging from 35% - 69% will be in moderate and scores greater than 70% will be considered as higher cooperation level.

Compliance of patient will be assessed by clinical compliance evaluation form (CCE) which comprises of four factors i.e. oral hygiene, maintenance of appliance, punctuality of appointments and appliance wear . These forms will be filled by co-investigator of the study. Each component has the same scores of 25, making total of 100. Calculation of patient's compliance on clinical compliance evaluation form will be the same as done by Richter et al. Maintenance of appliance, punctuality of appointments and appliance wear will be recorded from orthodontic record files while oral hygiene will be assessed when patient will come for their regular orthodontic visit. Presence of soft white plaque will be recorded on surface of bracket.

Compliance Check:

Two compliance log will be maintained one by the patient at home and other one by the primary investigator. A compliance log maintained by the primary investigator will be via telephone call to the participants in all groups to remind them to use the intervention. This phone call will be made to check whether the participants have used the intervention or not as instructed. If the participants have not used the intervention they will be requested to use the intervention and a final confirmation call will be made to check the compliance in few days again. Both the compliance log maintained by the patient at home and by the primary investigator will be compared to check the overall compliance of the participant at the end of the study.

After taking the baseline measurements by the investigator will unseal the envelope from Clinical Trials Unit (CTU), containing information regarding the intervention to be used on the participants based on randomization. The participants will be sent home and will be recalled for re-evaluation after every month till 3 months (T1,T2 and T3) The compliance will be assured by providing the log sheet to the participants . Additionally, after 2 weeks interval, all patients will be reminded by the investigator via phone call to check the compliance with the intervention.

Ethical considerations:

The study will be conducted according to the CONSORT guidelines and guidelines of World Medical Association's Declaration of Helsinki and the principles of GCP (Good Clinical Practice). All those patients who fulfilled the inclusion criteria will receive detailed information regarding the study and only those patients will be included who signed an informed consent. Any subsequent protocol amendments will be submitted to ERC and regulatory authorities for approval. The trial will be conducted in compliance with regulations, and a copy of interim analysis and final study report will be submitted to ERC.

Possible risks or benefits:

There are no known risks involved in this study as the study is based on communicating necessary information through video method and plaque disclosing tablets. Plaque disclosing tablets are considered to be safe for usage and are available as over the counter drugs. However, slight coloration of the mouth may last for more than 24 hours and stains on clothing as the coloring agent is strong. Benefits include finding the best modality to motivate orthodontic patients in improving oral hygiene during the course of the treatment.

Adverse events:

There is no adverse event reported in the literature related to the plaque disclosing tablets. The trial related events would be covered by the Department of Surgery. Slight discoloration of the oral tissues may last for up to 24 hours after using plaque disclosing tablets and stains on clothing can occur as the coloring agent are strong, these minor adverse events would be managed by prior counseling of the participants. These adverse events will be recorded and reported to ERC within a specified period of time, while no serious adverse event are expected.

Right of refusal to participate and withdrawal:

Participants will be given a choice to either participate or refuse to participate in the study. All participants non-compliant with using plaque disclosing tablets or watching the OHI video will be reinforced by phone calls, while comparing the compliance log sheets provided to them and other maintained by the PI.

Stopping rule:

The trial would be stopped if any of the intervention does not control plaque or if there is a deterioration of periodontal health as revealed by increasing GI, BI and OPI scores in the interim analysis done after recruiting 15 patients in each arm.

Incentive:

After one month (T1) all patients will be offered oral prophylaxis free of cost. If the indices are still high, and clinical examination shows a higher score of gingival inflammation, additional measures such as topical metronidazole gel and antibiotics will be given to control the gingival inflammation.

Patient confidentiality, access and storage:

The information provided by the participant will remain confidential. Nobody except the investigators will have access to it. Participants' name and identity will not be disclosed at any time. However, the data may be seen by ERC, DSMB or any local regulatory body. As per GCP and other guidelines, data will be retained for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing orthodontic treatment with fixed appliance (FAT) since 6 months
* Patients of both gender, aged 18-36 years. As, chances of declining periodontal status increases after 36 years of age.
* Patients having an Andriod phone with Whatsapp application installed..
* Patients with all bonded teeth mesial to the first molars.
* Healthy patients with no co-morbids such as rheumatic fever, blood dyscrasias, congenital heart disease or diabetes mellitus.
* Subjects with gingivitis as assessed by bleeding index (score ≤1), orthodontic plaque index (score ≤2) and gingival index (score ≤1) as assessed by Williams -Probe.
* All patients who will give consent for participation.

Exclusion Criteria:

* Subjects with clinical attachment loss of greater than 2 mm on two sites.
* Pregnant or lactating females.
* Subjects with removable/fixed dental prosthesis or banded teeth.
* History of surgical or nonsurgical periodontal therapy in the last 6 months.
* Current smokers or smokeless tobacco users. (According to glossary of Centers for Disease Control and Prevention, an adult who has smoked 100 cigarettes in his or her lifetime and who currently smokes cigarettes is considered to be current smoker).
* Patients having systemic reasons for periodontal diseases for example uncontrolled diabetes, hypertension.

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Gingival Index (GI) | 10 months
  0.No inflammation
  1. Mild inflammation: slight change in color, slight edema, no bleeding on probing
  2. Moderate inflammation: moderate glazing, redness, bleeding on probing
  3. Severe inflammation: marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding
Bleeding Index (BI): | 10 months
  0.Absence of bleeding after 30 seconds
  1. Bleeding observed after 30 seconds
  2. Immediate bleeding
Orthodontic Plaque Index (OPI) | 10 months
  0.No plaque deposits on the tooth surface surrounding the bracket base
  1. Plaque deposits on one tooth surface at the bracket base
  2. Plaque deposits on two tooth surfaces at the bracket base
  3. Plaque deposits on three tooth surfaces at the bracket base
  4. Plaque deposits on four tooth surfaces at the bracket base and/or gingival inflammation indicators (plaque deposits near the gingiva do not necessarily have to be present)

SECONDARY OUTCOMES:
Orthodontic Patient Cooperation Scale (OPCS) | 11 months
  1. This patient keeps appointments and is prompt. ( ) Always ( ) Frequently ( ) Sometimes ( ) Rarely ( ) Never
  2. This patient has distorted wires and/or loose bands. ( ) Always ( ) Frequently ( ) Sometimes ( ) Rarely ( ) Never
  3. This patient acts enthusiastic and interested in treatment. ( ) Always ( ) Frequently ( ) Sometimes ( ) Rarely ( ) Never
  4. This patient's behavior is sullen, hostile, belligerent, or rude. ( ) Always ( ) Frequently ( ) Sometimes ( ) Rarely ( ) Never
  5. This patient cooperates in the use of headgear and/or elastics. ( ) Always ( ) Frequently ( ) Sometimes ( ) Rarely ( ) Never
  6. This patient complains about treatment procedures. ( ) Always ( ) Frequently ( ) Sometimes ( ) Rarely ( ) Never
  7. This patient demonstrates excellent oral hygiene. ( ) Always ( ) Frequently ( ) Sometimes ( ) Rarely ( ) Never
  8. This patient complains about wear braces. ( ) Always ( ) Frequently ( ) Sometimes ( ) Rarely ( ) Never
Clinical compliance evaluation form (CCE) | 11
  Oral Hygiene:
  Plaque:
  RU6 RU1 LU6 LU1 RL6 LL6 None 4 4 4 4 4 4 Below bracket 3 3 3 3 3 3 On and below bracket 2 2 2 2 2 2 Above and below bracket 1 1 1 1 1 1
  Appointment Punctuality:
  On time or before 25 15-30 mins late 20 More than 30 mins late 15 Change Appointments in 24hrs 10 No Show 0
  Appliance Wear:
  Time HG Elastics 90-100% 25 25 80-90% 21 21 70-80% 18 18 60-70% 15 15 50-60% 12 12 40-50% 09 09 30-40% 06 06 20-30% 03 03 10-20% 0 0
  Appliance Maintenance:
  No breakage or bend in archwire 25 No breakage but mild bends in archwire 15 Moderate bends in archwire 10 Loose bands 5 Broken bracket or lose appliance 0 Scores Oral Hygiene:________________________ Appointment Punctuality:___________________ Appliance wear:________________________ Appliance maintenance:_________________________

CONTACTS AND LOCATIONS:
Overall Officials: Rashna Hoshang Sukhia, BDS, FCPS, Principal Investigator — Aga Khan University and Hospital
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF